CLINICAL TRIAL: NCT00761527
Title: Post-marketing Surveillance of the Safety, Tolerability and Efficacy of Desloratadine Syrup Among Filipino Pediatric Patients
Brief Title: Observation of Side Effects and Effectiveness of Desloratadine (Aerius) Syrup in Filipino Children (Study P05634)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P05634
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2012-03-01 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Seasonal; Rhinitis, Allergic, Perennial; Urticaria
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic, Perennial; Urticaria | interventions — desloratadine

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with allergic rhinitis or idiopathic urticaria: Outpatient pediatric participants (ages 6 months-11 years) in the Philippines with a diagnosis of allergic rhinitis or chronic idiopathic urticaria.
  Interventions: Drug: Desloratadine Syrup

INTERVENTIONS:
Drug: Desloratadine Syrup — Desloratadine (Aerius) Syrup;
  Dose selection was based upon the age of the participant, and the timing of dose for each participant was once daily (QD) as described in the Product Insert for 14 days:
  * Children 6 through 11 years of age, 5 mL (milliliters) of Aerius Syrup (2.5 mg [milligrams] of desloratadine)
  * Children 1 through 5 years of age, 2.5 mL of Aerius Syrup (1.25 mg of desloratadine)
  * Children 6 months to 11 months of age, 2 mL of Aerius Syrup (1 mg of desloratadine)
  Other Names: Aerius, Clarinex, SCH 34117, descarboethoxyloratadine

SUMMARY:
The purpose of this study is to observe the side effects of desloratadine syrup and how effective it is in relieving symptoms of allergic rhinitis or hives in Filipino children. The participants will take desloratadine syrup for 14 days. At the end of treatment, side effects will be recorded, as well as how the participants tolerate the medication. Effectiveness will also be rated at the end of treatment.

DETAILED DESCRIPTION:
Physicians who commonly prescribed desloratadine treatment as standard care of treatment were selected enroll participants.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient pediatric participants, male or female, aged 6 months to 11 years
* Diagnosis of allergic rhinitis or chronic idiopathic urticaria

Exclusion Criteria:

* Known hypersensitivity to desloratadine

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A total of 3000 prospective outpatient pediatric participants with either allergic rhinitis or chronic idiopathic urticaria will be enrolled in the study coming from about 300 sites in the Phillipines
Sampling Method: Non-Probability Sample
Enrollment: 2980 (Actual)
Dates: Start 2008-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The total number of participants enrolled was 2980. A total of 2978 participants received at least one dose of study medication.
Groups:
- Desloratadine (Aerius) Syrup: Pediatric participants with a diagnosis of allergic rhinitis or chronic idiopathic urticaria received Desloratadine (Aerius) Syrup. Dose selection was based upon the age of the participant, and the timing of dose for each participant was once daily (QD) as described in the Product Insert for 14 days:
  * Children 6 through 11 years of age, 5 mL (milliliters) of Aerius Syrup (2.5 mg [milligrams] of desloratadine)
  * Children 1 through 5 years of age, 2.5 mL of Aerius Syrup (1.25 mg of desloratadine)
  * Children 6 months to 11 months of age, 2 mL of Aerius Syrup (1 mg of desloratadine)
Period: Overall Study
Arm/Group | Desloratadine (Aerius) Syrup
Started | 2980
Received One Dose of Study Medication | 2978
Completed | 2958
Not Completed | 22
Not completed — Adverse Event | 3
Not completed — Poor Compliance | 8
Not completed — Lost to Follow-up | 9
Not completed — Unknown reason | 2

BASELINE CHARACTERISTICS:
Arm/Group | Desloratadine (Aerius) Syrup
Number analyzed (Participants) | 2978
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.74 (3.272)
Sex/Gender, Customized [Number; unit: Participants] — Number of participants with non-missing data for the relevant variable in the safety population (N= 2968) which included all participants who had taken at least one dose of study medication.
  Participants
    Male | 1511
    Female | 1457
    Missing Data | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events Reported By Category After 14 Days of Treatment
Description: Safety was assessed by determining the incidence of all Adverse Events (AE) which occurred between Baseline Visit (Day 1) & Final Visit (Day 15) & were recorded in Case Report Forms. Total number of AEs reported were presented in several categories. Classification, causality & intensity for AEs were determined by investigator after obtaining sufficient information. A Serious Adverse Event (SAE) was any adverse drug experience that resulted in: death; life-threatening condition; inpatient hospitalization/prolongation of existing hospitalization; persistent or significant disability/incapacity.
Time Frame: 15 Days
Population: The Safety population included all participants who had taken at least one dose of Desloratadine Syrup.
Measure: Number; unit: Adverse Events
Arm/Group | Desloratadine (Aerius) Syrup
Number analyzed (Participants) | 2978
Adverse Events
  Total Number of AEs | 26
  Number of Mild AEs | 21
  Number of Moderate AEs | 4
  Number of Severe AEs | 1
  Number of Treatment-related AEs | 20
  Number of Mild Treatment-related AEs | 19
  Number of Moderate Treatment-related AEs | 0
  Number of Severe Treatment-related AEs | 1
  Number of SAEs | 1
  Number of Treatment-related SAEs | 0

2. Primary Outcome: Safety of Desloratadine Syrup Reported by Number of Participants Experiencing Adverse Events After 14 Days of Treatment
Description: Safety was assessed by determining the incidence of all AEs which occurred between Baseline Visit (Day 1) & Final Visit (Day 15) & were recorded in Case Report Forms. Number of participants experiencing AEs were presented in several categories. Some AEs lead to discontinuation (d/c). Classification, causality & intensity for AEs were determined by investigator. A SAE was any adverse drug experience that resulted in any of the following: death; life-threatening condition; inpatient hospitalization/prolongation of existing hospitalization; persistent or significant disability/incapacity.
Time Frame: 15 Days
Population: The Safety population included all participants who had taken at least one dose of Desloratadine Syrup.
Measure: Number; unit: Participants
Arm/Group | Desloratadine (Aerius) Syrup
Number analyzed (Participants) | 2978
Participants
  Number of Participants with AEs | 24
  Number of Participants with Mild AEs | 21
  Number of Participants with Moderate AEs | 2
  Number of Participants with Severe AEs | 1
  Number of Participants with Treatment-related AEs | 20
  Number of Participants with AEs - Temporary d/c | 1
  Number of Participants with AEs - Permanent d/c | 2
  Number of Participants with AEs - Withdrawal | 2
  Number of Participants with SAEs | 1
  Number of Participants with Treatment-related SAEs | 0
  Number of Participants Who Died Due to AEs | 0

3. Secondary Outcome: Investigator Assessment of Clinical Efficacy
Description: Investigator assessment of clinical efficacy of Desloratadine Syrup in relieving participants' symptoms of either allergic rhinitis or chronic idiopathic urticaria at final visit (Day 15). The number of participants categorized by investigator as: improved, no improvement, or worsened was reported at Day 15.
Time Frame: Day 15
Population: ITT Population, which consisted of all participants who had taken at least one dose of Desloratadine Syrup and had a post baseline clinical efficacy assessment (N=2956). For 4 participants, a clinical efficacy assessment was not reported.
Measure: Number; unit: Participants
Arm/Group | Desloratadine (Aerius) Syrup
Number analyzed (Participants) | 2952
Participants
  Improvement | 2913
  No Improvement | 39
  Worsened | 0

4. Primary Outcome: Participant Global Tolerability Assessment
Description: The participant's global assessment of tolerability with the medication was assessed using a categorical scale as follows:
  * Excellent
  * Very Good
  * Good
  * Fair
  * poor
  Parent or guardian of each participant followed up for a final visit after 14 days (Day 15) at which tolerability was rated and reported for entire treatment period. Number of participants in each category is presented.
Time Frame: Day 15
Population: The Safety population included all participants who had taken at least one dose of Desloratadine Syrup (N=2978). For 31 participants, tolerability was not assessed.
Measure: Number; unit: Participants
Arm/Group | Desloratadine (Aerius) Syrup
Number analyzed (Participants) | 2947
Participants
  Excellent | 1278
  Very Good | 1339
  Good | 307
  Fair | 15
  Poor | 8

ADVERSE EVENTS:
Time Frame: Safety Population included all participants who had taken at least one dose of Desloratadine Syrup.
Arm/Group | Desloratadine (Aerius) Syrup
Serious Adverse Events (participants affected / at risk) | 1/2978
Other Adverse Events (participants affected / at risk) | 0/2978
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desloratadine (Aerius) Syrup (N=2978)
Pneumonia (Infections and infestations) | 1 (1) — Reported by the prescribing physician as unrelated to study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
SPONSOR is the owner of all the data in the record forms including subsequent reports relating to this study. The prescribing physicians & investigators agree only to use such information to conduct the study & will not be able to publish the results of any part of this study without previous written authorization from SPONSOR. By signing the protocol, the investigator accepts that the results may be used in written publications & for the purpose of providing information to health professionals.